CLINICAL TRIAL: NCT03029338
Title: CD19 CAR T Cells in Patients With Relapsed or Refractory CD19 Positive B-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QT2016003
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2022-01

CONDITIONS: Lymphomas Non-Hodgkin's B-Cell; Relapse
Keywords: lymphoma; non-hodgkin; B-cell; CD19 CAR T cells; refractory; relapse
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence; Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 CAR T cells (Experimental): CD19 CAR T cells will be intravenously infused to patient in a three-day split-dose regimen: 10% on day 0, 30% on day 1 and 60% on day 2.
  Interventions: Biological: CD19 CAR T cells

INTERVENTIONS:
Biological: CD19 CAR T cells — CD19 CAR T cells was transduced with a lentiviral vector to express anti-CD19 scFv TCRζ:4-1BB.

SUMMARY:
In this single-center, open-label, no control, prospective clinical trial, a total of 10 relapsed or refractory CD19 positive B-cell Non-Hodgkin Lymphoma (NHL) patients will be enrolled.CD19 CAR T cells(total dose of 2×10^6/kg-1×10^7/kg) will be intravenously infused to patient in a three-day split-dose regimen: 10% on day 0, 30% on day 1 and 60% on day 2. The purpose of current study is to determine the clinical efficacy and safety of CD19 CAR T cells in patients with relapsed or refractory CD19 positive B-cell lymphoma.

DETAILED DESCRIPTION:
In this single-center, open-label, nonrandomized, no control, prospective clinical trial, a total of 10 relapsed or refractory CD19+ B-cell Non-Hodgkin Lymphoma (NHL) patients will be enrolled. CD19 CAR T cells transduced with a lentiviral vector to express anti-CD19 scFv TCRζ:4-1BB, will be administered by i.v. injection in a three-day split-dose regimen: 10% on day 0, 30% on day 1 and 60% on day 2. Side effects of CD19 CAR T cells therapy will be monitored. The purpose of current study is to determine the clinical efficacy and safety of CD19 CAR T cells therapy in patients with relapsed or refractory CD19 positive B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 70 years with relapsed or refractory CD19 positive B-cell lymphoma.
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
* Adequate end organ function as defined by: Total bilirubin ≤ 1.5 x upper limit of normal（ULN）; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN; Creatinine ≤ 1.5 x ULN or any serum creatinine level associated with a measured or calculated creatinine clearance of ≥ 40ml/min.
* Male and female of reproductive potential must agree to use birth control during the study and for at least 6 weeks post study.
* Patients should sign informed consent form.

Exclusion Criteria:

* Patients with central nervous system involvement by lymphoma.
* Prior chemotherapy within 2 weeks before enrollment with the following exceptions: steroids, hydroxyurea, oral mercaptopurine, methotrexate, vincristine and thioguanine are permitted within 2 weeks of enrollment as maintenance or to reduce tumor load.
* Prior allogeneic hematopoietic stem cell transplant (HSCT) ≤ 4 months before enrollment. Patients must have completed immunosuppression therapy prior to enrollment. At enrollment, patients must not have≥ grade 2 acute GVHD, or either moderate or severe limited chronic GVHD, or extensive GVHD of any severity.
* Known systemic vasculitides, primary or secondary immunodeficiency(such as HIV infection or severe inflammatory disease).
* Major surgery within 4 weeks before enrollment.
* Impaired cardiac function:Ejection fraction ≤45 % on MUGA scan. QTc interval > 450msecs on baseline ECG. Myocardial infarction within 6 months prior to starting study; other clinically significant heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension, uncontrolled arrhythmias).
* Administration of live vaccine ≤ 4 weeks before enrollment.
* Other concurrent severe and/or uncontrolled medical conditions: Patients with another primary malignant disease, except those that do not currently require treatment; acute or chronic liver, pancreatic or severe renal disease; another severe and/or life-threatening medical disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 2 years

SECONDARY OUTCOMES:
Severity of the adverse events | 2 years
Response rate | 12 months
Progression-free survival(PFS) | 2 years
Persistence of CAR T cells in vivo | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dehui Zou, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu W, Xie T, Zhang Z, Huang W, Liu H, Sui W, Deng S, Lv R, Wang Y, Wang Q, Xiong W, Xu Y, Lv L, Ma Y, Qiu L, Wang J, Zou D. Long-term outcomes of CNCT19 chimeric antigen receptor T-cell therapy in relapsed or refractory aggressive B-cell lymphoma. Chin Med J (Engl). 2025 Sep 17. doi: 10.1097/CM9.0000000000003716. Online ahead of print. PMID 40960310